CLINICAL TRIAL: NCT06569433
Title: Efficacy of Therapeutic Exercise Compared to Femoral Nerve Mobilisation in Knee Tendinosis: Randomised Clinical Trial
Brief Title: Efficacy of Therapeutic Exercise Compared to Femoral Nerve Mobilisation in Knee Tendinosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Silvia Martinez, Investigador principal, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Silvia M
Record Dates: First submitted 2024-08-11; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Chronic Patellar Tendinopathy
MeSH Terms: interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: The following criteria for inclusion and exclusion of participants have been established:
  Inclusion criteria:
  * Patients aged between 18 and 40 years.
  * Patients with chronic or acute knee tendinosis.
  * Patients with pain or functional limitation
  Exclusion criteria:
  * Patients with any contraindication to treatment.
  * Patients with a history of recent knee surgery or serious injury
  * Who present neurological pathologies
  * Who are using other physiotherapy techniques
  Prior to registration each participant must undergo a physical assessment, including a medical history check and provide information on neurological and trauma pathologies. Those who meet the criteria will be assigned to one of the two study groups.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic exercise (Active Comparator): In the interventions, the control group performing therapeutic exercise only, will perform a specific exercise programme for knee tendinitis under the supervision of a physiotherapist,
  Interventions: Procedure: THERAPEUTIC EXERCISE AND MOBILISATION OF THE FEMORAL NERVE
- Femoral nerve movilization (Active Comparator): will receive therapeutic exercise sessions and femoral nerve mobilisations performed by a trained physiotherapist.
  Interventions: Procedure: THERAPEUTIC EXERCISE AND MOBILISATION OF THE FEMORAL NERVE

INTERVENTIONS:
Procedure: THERAPEUTIC EXERCISE AND MOBILISATION OF THE FEMORAL NERVE — the control group that will perform only therapeutic exercise will perform a specific exercise programme for knee tendinitis under the supervision of a physiotherapist, while the intervention group that will perform therapeutic exercise plus femoral nerve mobilisation will receive therapeutic exercise sessions and femoral nerve mobilisations performed by a trained physiotherapist.
  The intervention will last for 6 weeks, during which 60-minute sessions will be held at the centre, measurements will be taken during the six weeks, using standardised questionnaires to evaluate the variables (set out below) and always measuring the range of movement and femoral nerve mobility with the Slump Test on the same day of the week and at the same time of treatment.

SUMMARY:
Tendons, located between muscle and bone, transmit force from the former to the latter, allowing joint movement. They are composed mainly of collagen, elastin and water, and are divided into three zones: osteotendinous junction (tendon-bone), myotendinous junction (muscle-tendon) and the tendon body.

Knee tendinosis is a pathology that affects the tendons of this joint due to the breakdown of collagen in the tendon body, characterised by pain during and after exercise, inflammation and loss of function. It is common in athletes, especially in jumping sports such as basketball and volleyball, due to repetitive strain, injury or ageing. Factors such as weight, leg length and muscle strength can influence its development. Radiologically, patellar tendon thickening, and abnormalities are seen.

Treatment includes eccentric exercises, shock wave therapy, ultrasound-guided sclerosis, anti-inflammatory drugs, plasma injections and aprotinin. Neurodynamic theory suggests that altered mechanosensitivity of the femoral nerve may contribute to knee pain, and neurodynamic techniques can improve nerve mobility and reduce symptoms.

A strength exercise with isometric contractions can decrease pain for up to 45 minutes, being a therapeutic option for patellar tendinopathy without affecting muscle strength.

The research project presented in the master's thesis aims to compare the effectiveness of femoral nerve mobilisation and therapeutic exercise in the treatment of knee tendinosis.

DETAILED DESCRIPTION:
Nowadays, tendon injuries affect a large part of the population, especially people who practice sports and the working population in industrial sectors, although they have also been observed in sedentary people. In terms of occupational diseases, these injuries account for more than 35% in the most industrialised countries of the European Union.

The indirect costs of tendinopathies can be significant in terms of lost productivity and workers' compensation.

Despite the lack of specific data on the economic impact of knee tendinosis on society, given the high prevalence of this condition, it is crucial to study its treatment to reduce recovery time and associated costs. Both therapeutic exercise and femoral nerve mobilisation are supported by scientific evidence suggesting their efficacy in the treatment of knee tendinitis. However, it is important to specifically investigate and compare how these interventions affect symptoms and function in patients with this condition.

Therapeutic exercise prevents injury and aids in the regeneration of the knee extensor system. The goal is to restore adequate strength, flexibility and endurance, as well as to correct joint limitations.

It has been studied that the success of treatment of tendinopathies may be determined by the adaptation of the exercise loads to the capacity of the tendons.

ELIGIBILITY:
Inclusion Criteria:

* - Patients aged 18 to 40 years old
* Patients with chronic or acute knee tendinosis
* Who have pain or functional limitation

Exclusion Criteria:

* Patients with a contraindication to treatment
* Patients with a history of recent knee surgery or serious injury
* Who present neurological pathologies
* Who are using other physiotherapy techniques

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-20 (Estimated); Primary Completion 2024-09-20 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
The 'pain' variable | 6 weeks
  The variable 'pain' is subjective and qualitative and is measured quantitatively to facilitate its analysis. In this case the Visual Analogue Scale (VAS) will be used, which facilitates the subjective evaluation of the intensity of the pain that the patient experiences, through a score based on their perception of pain, It ranges from 0 (being the lowest score therefore there is no pain) to 10 (being the highest score therefore it is at its maximum pain level)
functionality (VISA-P questionnaire) | 6 weeks
  the VISA-P questionnaire which allows us to classify tendinopathy according to the severity of the symptoms and the functional capacity of the patients.

IPD SHARING:
Plan to Share IPD: No